CLINICAL TRIAL: NCT04180358
Title: Capacity Builders Inc. Navajo Youth Builders Personal Responsibility Education Innovation Strategies Project Effectively Educating Navajo Youth on the Prevention of Adolescent Pregnancy, Sexually Transmitted Infections, and HIV/AIDS
Brief Title: Capacity Builders Inc. Navajo Youth Builders Personal Responsibility Education Innovation Strategies Project
Acronym: PREIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capacity Builders Inc. (Other)
Collaborators: Mathematica Policy Research, Inc. (Other); Family and Youth Services Bureau (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 90AP2687-01-00; 90AP2687-00 (Other Grant/Funding Number: Family and Youth Services Bureau)
Record Dates: First submitted 2019-11-22; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Sexual Abstinence; Responsible Sex
Keywords: Navajo; Sex; Abstain; Culture; Random; Control; Trial; PREIS
MeSH Terms: conditions — Sexual Abstinence; Safe Sex; Coitus

STUDY DESIGN:
Intervention Model Description: CBI will implement the Youth Builders PREIS Native STAND curriculum, a comprehensive sexual health curriculum designed for Native high school students that focuses on STI's, HIV/AIDS, and teen pregnancy prevention and covers drug and alcohol use, suicide, and dating violence. Twenty-seven sessions support healthy decision-making through interactive discussions and activities that promote diversity, self-esteem, goals and values, team building, negotiation and refusal skills, and effective communication. Youth Build will enroll 834 youth in 3 cohorts with 42 clusters of 20 students, each who will be randomly assigned to an impact or a comparison group. Students will complete pre and post survey questionnaires and be provided incentives to maintain program participation. The program will have 4 staff: Project Director, Project Coordinator, and 2 Prevention Educations responsible for collecting data and tracking progress as well as implementing the curriculum
Who Masked: Participant
Masking Description: The impact group who is randomly selected will receive the intervention in Physical Education and Health Education classes. The control group will receive the general health and physical education curriculum provided by New Mexico's Public Education Department. No students will take a class twice unless there is a failing grade. Student will be tracked throughout the school year to ensure there is no cross contamination. Additionally, Counselors will work closely with Capacity Builder's program staff to ensure that in between semesters, students will remain in their original group. Program staff will double check at the beginning of each semester to crosswalk student assignments. Additionally, participants in the past Capacity Builder's Inc. Teen Pregnancy Prevention programs will be excluded to minimize the risk that the comparison group participants are exposed to teen pregnancy prevention curricula and, thus, to increase contrast between the intervention and control conditions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impact group (Experimental): The impact group will receive the interventions in the classrooms
  Interventions: Behavioral: Native STAND
- Comparison group (Placebo Comparator): Comparison group will not receive the intervention
  Interventions: Behavioral: Regular Health/Physical Education Curriculum

INTERVENTIONS:
Behavioral: Native STAND — Native STAND is a comprehensive sexual health curriculum for Native high school students that focuses on sexually transmitted infections, HIV/AIDS, and teen pregnancy prevention, while also covering drug and alcohol use, suicide, and dating violence. Twenty-seven sessions support healthy decision-making through interactive discussions and activities that promote diversity, self-esteem, goals and values, team building, negotiation and refusal skills, and effective communication. Sessions will be conducted in regular Physical Education and/or Health Education classes during classroom/school hours.
  Arms: Impact group
Behavioral: Regular Health/Physical Education Curriculum — General health and physical education curriculum provided by New Mexico's Public Education Department.
  Arms: Comparison group

SUMMARY:
Capacity Builders (CBI) will implement the Youth Builders PREIS curriculum Native Students Together Against Negative Decisions (Native STAND) which aims to reduce pregnancies, births, and sexually transmitted infections (STI's) including HIV/AIDS among high-risk youth populations by implementing culturally sensitive curriculum based on Navajo positive youth development. The study has two hypotheses: (1) Do students assigned to the Youth Builders program have a greater chance of abstaining from sexual activity (i.e. oral, vaginal and anal) in the last 3 months as compared to students assigned to the comparison group, measured at 12 month and 18 month follow up? (No vaginal sexual intercourse, report abstinence at 12 and 18 random assignment month follow up); (2) Do students assigned to the Youth Builders program have a greater change of abstaining from sex or practicing safe sex (i.e. using a male or female condom, or other means of birth control if they have sex), than students assigned to the comparison group, measured at 12 and 18 months after random assignment? (No sexual activity or use contraception if engage in sex at 12 month and 18 month follow up.

DETAILED DESCRIPTION:
Capacity Builders (CBI) will implement the Youth Builders PREIS curriculum Native STAND, recruiting Navajo youth in grades 9-11 and between the ages 14-18 who attend school in the Consolidated School District in New Mexico. Using the Theory of Reasoned Action as a theoretical framework, the curriculum will be administered in classrooms over 27 sessions lasting 45 minutes. The curriculum will entail lessons conducted in either Physical Education or Health Classes and youth will be randomly assigned to two groups by the local program evaluator. Youth will be required to obtain signed consent and assent forms prior to participating in the intervention program. Youth will complete pre and post surveys to measure program outcomes. Random assignment will be conducted for the impact and comparison groups by being placed into a pool; students will be blindly pulled to become the impact group. Groups will be stratified to ensure balance between treatment and comparison groups. Quarterly evaluation reports (QERs) and an annual evaluation report will be provided to the Action Team for review.

Capacity Builder's Inc. (CBI) Youth Builders PREIS program seeks to test a modification of the Native STAND curriculum in Northwest New Mexico with at least 834 Navajo teens and 3 cohorts. The curriculum is intended to reduce pregnancies, births, and STI's including HIV/AIDS among high-risk youth populations by implementing culturally sensitive curriculum based on Navajo positive youth development. Additional curriculum of adulthood preparation subjects will increase participant knowledge in the areas of: healthy relationships, adolescent development, communication skills, healthy life skills. Youth Builders will be delivered within the traditional school day, embedded into regularly scheduled learning time. Presented once each week for 27 weeks over a 36-week school year, Youth Builders will reach students where they are, overcoming many challenges associated with retention. The project will support a Randomized Controlled Experimental Design. CBI will create valuable resources to support Youth Builders replication nationwide, including a comprehensive Youth Builders Blueprint, describing all action steps taken to achieve goals and objectives. In addition to action steps, the Youth Builders Blueprint will include: program curriculum; curricular map; training materials; sample parent consent forms; sample referral procedures / policies; staff training schedules; sample partnership agreements; Action Team meeting minutes,QERs, and annual evaluation reports The Youth Builders Blueprint will be available in both print and online format, and will be widely disseminated throughout the CBI network of non-profit agencies, Tribes, and school districts across the United States. Conference presentation will be ongoing at state and national conferences.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 14-18
* In grades 9-11
* Provide parental consent and participant assent to participate in the study
* Students in the first two groups will be allowed to participate in the intervention if they are enrolled in the classroom that will be receiving the intervention
* Students in the third group will be allowed to participate in the intervention only if they were part of the study's intervention group

Exclusion Criteria:

* Not have previously participated in any of the following past CBI Teen Pregnancy

Prevention programs:

* New Mexico's Department of Health - Wyman's Teen Outreach Program
* Success with Adolescent Goals, inclusive of the Above the Waist Curriculum
* Students in 12th grade
* Study participants from previous cohorts

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 834 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-09-29 (Estimated)

PRIMARY OUTCOMES:
Abstaining from sexual activity | pre test, post test after 27 lessons, short term follow up at 12 months, long term follow up at 18 months
  Do students assigned to the Youth Builders program have a greater chance of abstaining from sexual activity (i.e. oral, vaginal and anal) in the last 3 months compared to students assigned to the comparison group at 12 month follow up and 18 month follow up? (No vaginal sexual intercourse, report abstinence at 12 and 18 random assignment month follow up?
Abstaining from sex or practicing safe sex | pre test, post test after 27 lessons, short term follow up at 12 months, long term follow up at 18 months
  Do students assigned to the Youth Builders program have a greater chance of abstaining from sex or practicing safe sex (i.e. using a male or female condom, or other means of birth control if they have sex), than students assigned to the comparison group at 12 month follow up and 18 month follow up? (No sexual activity or use contraception if engage in sex at 12 and 18 month follow up)?

SECONDARY OUTCOMES:
Positive impact on participants' assertive communication/negotiation skills | pre test, post test after 27 lessons, short term follow up at 12 months, long term follow up at 18 months
  To what degree does the Youth Builders curriculum have a positive impact on participants' assertive communication/negotiation skills?
Positive impact on the peer to peer communication/discussing expectations habits of participants | pre test, post test after 27 lessons, short term follow up at 12 months, long term follow up at 18 months
  To what degree does the Youth Builders curriculum have a positive impact on the peer to peer communication/discussing expectations habits of participants?
Positive impact on the family communication/discussing expectations habits of participants | pre test, post test after 27 lessons, short term follow up at 12 months, long term follow up at 18 months
  To what degree does the Youth Builders curriculum have a positive impact on the family communication/discussing expectations habits of participants?

OTHER OUTCOMES:
Greater chance of not becoming (female) or getting (male) the opposite sex pregnant, than students assigned to the comparison group at 12 and 18 months after random assignment | pre test, post test after 27 lessons, short term follow up at 12 months, long term follow up at 18 months
  Do students assigned to the Youth Builders program have a greater chance of not becoming (female) or getting (male) the opposite sex pregnant, than students assigned to the comparison group at 12 and 18 months after random assignment?

CONTACTS AND LOCATIONS:
Overall Officials: Lois Ritter, Principal Investigator — Capacity Builders Inc.
Locations (1):
- Capacity Builders Inc., Farmington, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Healthy Native Youth — http://www.healthynativeyouth.org/
- See also: Native STAND (Students Together Against Negative Decisions) — http://www.nativestand.com/
- See also: Capacity Builders — http://capacitybuilders.info/
- See also: Navajo Nation Human Research Review Board — http://www.nnhrrb.navajo-nsn.gov/